CLINICAL TRIAL: NCT06537960
Title: Intérêt Des Images Tardives Pour le Bilan d'Extensions en TEP-TDM au 18FGD Des Cancers de Vessie Infiltrant le Muscle (TARDITEP)
Brief Title: Interest of Late Images for the Assessment of Extensions in 18FGD PET-CT of Muscle-Invasive Bladder Cancers
Acronym: TARDITEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021_0151
Record Dates: First submitted 2024-07-30; First posted 2024-08-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18FDG PET-CT (Other): 18FDG PET-CT will be performed in 2 phases:
  1. st standard phase: Standard acquisition (vertex to mid-thigh) at 1 hour post-injection of radiotracer
  2. nd phase: Complementary abdomino-pelvic acquisition at 2.5 hours post radiotracer injection.
  Interventions: Procedure: 18FDG PET-CT

INTERVENTIONS:
Procedure: 18FDG PET-CT — 18FDG PET-CT will be performed in 2 phases:
  1. st standard phase: Standard acquisition (vertex to mid-thigh) at 1 hour post-injection of radiotracer
  2. nd phase: Complementary abdomino-pelvic acquisition at 2.5 hours post radiotracer injection.

SUMMARY:
The goal of this study is to demonstrate a significant gain in sensitivity versus surgical curage (extended pelvic) for initial lymph node staging of late FDG-PET images (2.5 hours) versus standard images (1 hour), analyzed by side (right iliac/left iliac areas in Patients with muscle-invasive bladder tumor (MIBT) (≥pT2) referred for FDG-PET in the nuclear medicine department of Hôpital Foch as part of their initial extension workup.

Before performing 18FDG PET-CT, the operator checks that the patient has fasted for at least 6 hours and that blood glucose levels are below 11 mmol/l. In the absence of contraindication, intravenous (IV) injection of the radiopharmaceutical (18FDG at a dose of 3 MBq/kg) and a diuretic (Furosemide 20mg) will be performed as part of routine care. The 18FDG PET-CT scan will be performed in 2 phases:

1st phase: Standard acquisition (vertex to mid-thigh) at 1 hour post-injection of radiotracer. PET acquisition is coupled to a "base-dose" CT scan in spontaneous contrast, for anatomical location, measurement of lymph node size, and creation of an attenuation map, necessary for correction of attenuation and diffusion on PET images (DLP estimated at around 500 mGy.cm on average). Micturition is performed as part of routine care just before the first acquisition.

Phase 2: Complementary abdomino-pelvic acquisition at 2.5 hours post-injection (2 or 3 steps depending on patient size. This second PET acquisition is coupled to an "ultra-base-dose" CT scan in spontaneous contrast, to be used only for attenuation and diffusion correction (DLP estimated at around 100 mGy.cm on average). Micturition is performed 30 minutes before the second acquisition.

The patient's proposed therapeutic management will be decided at the PCR once the extension work-up has been carried out, as part of routine care. For this purpose, only "standard" 18FDG PET-CT images may be used.

As a general rule, patients with distant metastases (stage pT2N+M+) will receive palliative treatment, while surgical treatment from the outset, or after chemotherapy for patients with stage pT2N0M0 or pT2N+M0, will be discussed on a case-by-case basis at the multidisciplinary consultation meeting.

Late" images will be used after lymph node curage, in patients who have not had chemotherapy prior to surgery (cystectomy + extended pelvic lymph node curage), to determine the sensitivity of these complementary images.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older,
* With histologically proven muscle-invasive bladder cancer (≥pT2) at endoscopic bladder resection,
* Scheduled to undergo 18FDG PET-CT in the nuclear medicine department at Hôpital Foch,
* Having signed a consent form,
* Affiliated to a health insurance scheme.

Exclusion Criteria:

* Patient with a history of pelvic or genitourinary cancer,
* Patient with known metastatic disease,
* Patient with a contraindication to 18FDG PET-CT,
* Pregnant or breast-feeding woman,
* Patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity versus lymph node curage (per side) | 39 months
  Sensitivity versus lymph node curage (per side) for a blinded visual analysis, by two experts, with joint rereading in the event of discordance, of the two sets of images (1h and 2h30 post-injection), in patients who have not had chemotherapy prior to surgery (cystectomy + extensive pelvic lymph node curage).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France